CLINICAL TRIAL: NCT04635579
Title: Personalized Blood Flow Restriction for Anterior Cruciate Ligament Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Scott Telfer, EngD, Assistant Professor: School of Medicine, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00004543; 5P30AR072572-02 (NIH)
Record Dates: First submitted 2020-11-02; First posted 2020-11-19 (Actual); Results first posted 2022-02-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Anterior Cruciate Ligament Tear
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Anterior cruciate ligament reconstruction group (Experimental): Single session blood flow restriction of lower limb to individuals who have undergone anterior ligament reconstruction surgery
  Interventions: Device: Blood flow restriction
- Control group (Active Comparator): Single session blood flow restriction of lower limb to individuals who have no musculoskeletal injuries
  Interventions: Device: Blood flow restriction

INTERVENTIONS:
Device: Blood flow restriction — Intervention restricts blood flow to the lower limb as a percentage of the limb occlusion pressure

SUMMARY:
This is a cross-sectional study on the use of personalized blood flow restriction during rehabilitation exercises and its effects on biomechanics on people who have had an anterior cruciate ligament reconstruction and healthy controls

DETAILED DESCRIPTION:
Rehabilitation after surgical reconstruction of the anterior cruciate ligament (ACL) aims to reestablish the function of the knee. However, regaining previous levels of strength is challenging, with long-term muscle weakness frequently reported and thought to play a key role in the increased risk of knee osteoarthritis for individuals with a history of ACL damage. Effectively building muscle strength requires exercises with high resistance loads, however the joint stress and risk of further injury makes these types of activities inappropriate and unsafe for those rehabilitating after ACL reconstruction surgery and other injuries. Personalized blood flow restriction (BFR) training is a technique where the blood flow to the muscles being exercised is controlled by a pressure cuff to a predefined level, and has been shown to increase strength while exercising with significantly lower loads. Early results have been promising, however the effects of BFR on the biomechanics of the exercise as well as the acceptability in the ACL reconstruction population have not been explored. In this application, we propose a cross-sectional study designed to test the acceptability of BFR training for those undergoing rehabilitation from ACL reconstruction surgery and healthy controls during free standing exercises. We will also investigate the biomechanical effects of this rehabilitation technique. This application is part of a larger program of musculoskeletal research in this area being developed by the team. The results from the proposed project will inform the design of a clinical trial of personalized BFR after ACL reconstruction.

ELIGIBILITY:
Inclusion Criteria (ACL-R group):

* Must be undergoing rehabilitation for anterior cruciate ligament reconstruction surgery
* Must be at least 3 months post surgery.
* Attending clinician should confirm that they are able to take part in the trial

Exclusion Criteria:

* Any other orthopaedic, neurological, or other condition within the last 12 months that would affect ability to carry out the required exercises
* Any medical conditions that may affect circulation including, but not limited to, deep vein thrombosis, high blood pressure, and cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Telfer, EngD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available to researchers on request. Dataset includes all kinematic, kinetic and patient reported data.
Supporting Information: Study Protocol, Analytic Code
Time Frame: 11/19/2021 - 11/18/2026

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anterior Cruciate Ligament Reconstruction Group | Control Group
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anterior Cruciate Ligament Reconstruction Group | Control Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Full Range); unit: years] | 30.6 [21 to 50] | 28 [19 to 48] | 29.3 [19 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 8 | 9 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 17 | 18 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Knee Flexion
Description: Maximum difference in flexion motion of knee while performing exercise between baseline and blood flow restriction condition. Measured in degrees
Time Frame: 6 minutes
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Anterior Cruciate Ligament Reconstruction Group | Control Group
Number analyzed (Participants) | 20 | 20
Degrees | -0.05 (2.0) | 0.01 (5.14)

2. Primary Outcome: Knee Internal Rotation
Description: Maximum difference in internal rotation of knee while performing exercise between baseline and blood flow restriction condition. Measured in degrees
Time Frame: 6 minutes
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Anterior Cruciate Ligament Reconstruction Group | Control Group
Number analyzed (Participants) | 20 | 20
Degrees | 1.19 (1.4) | -0.03 (1.97)

3. Primary Outcome: Knee Varus
Description: Maximum difference in varus motion of knee while performing exercise between baseline and blood flow restriction condition. Measured in degrees
Time Frame: 6 minutes
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Anterior Cruciate Ligament Reconstruction Group | Control Group
Number analyzed (Participants) | 20 | 20
Degrees | 0.12 (1.25) | -0.36 (2.61)

4. Primary Outcome: Hip Flexion
Description: Maximum difference in flexion motion of hip while performing exercise between baseline and blood flow restriction condition. Measured in degrees
Time Frame: 6 minutes
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Anterior Cruciate Ligament Reconstruction Group | Control Group
Number analyzed (Participants) | 20 | 20
Degrees | -1.73 (2.27) | -2.9 (8.15)

5. Primary Outcome: Hip Adduction
Description: Maximum difference in adduction motion of hip while performing exercise between baseline and blood flow restriction condition. Measured in degrees
Time Frame: 6 minutes
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Anterior Cruciate Ligament Reconstruction Group | Control Group
Number analyzed (Participants) | 20 | 20
Degrees | 0.61 (1.9) | 1.52 (2.6)

6. Primary Outcome: Hip Internal Rotation
Description: Maximum difference in internal rotation motion of hip while performing exercise between baseline and blood flow restriction condition. Measured in degrees
Time Frame: 6 minutes
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Anterior Cruciate Ligament Reconstruction Group | Control Group
Number analyzed (Participants) | 20 | 20
Degrees | 1.49 (2.37) | 1.05 (2.6)

7. Primary Outcome: Knee Extension Moment
Description: Maximum difference in extension moment of knee while performing exercise between baseline and blood flow restriction condition. Measured in Newton meters per kilogram
Time Frame: 6 minutes
Measure: Mean (Standard Deviation); unit: Newton meters per kilogram
Arm/Group | Anterior Cruciate Ligament Reconstruction Group | Control Group
Number analyzed (Participants) | 20 | 20
Newton meters per kilogram | 0.31 (0.21) | 0.6 (0.26)

8. Primary Outcome: Knee Internal Rotation Moment
Description: Maximum difference in internal rotation moment of knee while performing exercise between baseline and blood flow restriction condition. Measured in Newton meters per kilogram
Time Frame: 6 minutes
Measure: Mean (Standard Deviation); unit: Newton meters per kilogram
Arm/Group | Anterior Cruciate Ligament Reconstruction Group | Control Group
Number analyzed (Participants) | 20 | 20
Newton meters per kilogram | -0.01 (0.05) | -0.02 (0.07)

9. Primary Outcome: Knee Adduction Moment
Description: Maximum difference in adduction moment of knee while performing exercise between baseline and blood flow restriction condition. Measured in Newton meters per kilogram
Time Frame: 6 minutes
Measure: Mean (Standard Deviation); unit: Newton meters per kilogram
Arm/Group | Anterior Cruciate Ligament Reconstruction Group | Control Group
Number analyzed (Participants) | 20 | 20
Newton meters per kilogram | 0.06 (0.05) | 0.12 (0.07)

10. Primary Outcome: Hip Extension Moment
Description: Maximum difference in extension moment of hip while performing exercise between baseline and blood flow restriction condition. Measured in Newton meters per kilogram.
Time Frame: 6 minutes
Measure: Mean (Standard Deviation); unit: Newton meters per kilogram
Arm/Group | Anterior Cruciate Ligament Reconstruction Group | Control Group
Number analyzed (Participants) | 20 | 20
Newton meters per kilogram | 0.09 (0.16) | 0.2 (0.14)

11. Primary Outcome: Hip Adduction Moment
Description: Maximum difference in adduction moment of hip while performing exercise between baseline and blood flow restriction condition. Measured in Newton meters per kilogram
Time Frame: 6 minutes
Measure: Mean (Standard Deviation); unit: Newton meters per kilogram
Arm/Group | Anterior Cruciate Ligament Reconstruction Group | Control Group
Number analyzed (Participants) | 20 | 20
Newton meters per kilogram | -0.01 (0.1) | -0.07 (0.14)

12. Primary Outcome: Hip Internal Rotation Moment
Description: Maximum difference in internal rotation moment of hip while performing exercise between baseline and blood flow restriction condition. Measured in Newton meters per kilogram
Time Frame: 6 minutes
Measure: Mean (Standard Deviation); unit: Newton meters per kilogram
Arm/Group | Anterior Cruciate Ligament Reconstruction Group | Control Group
Number analyzed (Participants) | 20 | 20
Newton meters per kilogram | -0.02 (0.13) | 0.05 (0.05)

13. Secondary Outcome: Exercise Difficulty Score
Description: Numerical Analogue Scale, 0-10, higher scores indicate greater difficulty
Time Frame: 6 minutes
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Anterior Cruciate Ligament Reconstruction Group | Control Group
Number analyzed (Participants) | 20 | 20
units on a scale | 4.0 [3 to 5.5] | 5.0 [4.5 to 6]

14. Secondary Outcome: Exercise Discomfort Score
Description: Numerical Analogue Scale, 0-10, higher scores indicate greater discomfort
Time Frame: 6 minutes
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Anterior Cruciate Ligament Reconstruction Group | Control Group
Number analyzed (Participants) | 20 | 20
units on a scale | 4.0 [3.5 to 5.5] | 4.5 [3 to 5]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Anterior Cruciate Ligament Reconstruction Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-04-24): https://cdn.clinicaltrials.gov/large-docs/79/NCT04635579/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-24): https://cdn.clinicaltrials.gov/large-docs/79/NCT04635579/SAP_001.pdf
  • Informed Consent Form (2018-04-24): https://cdn.clinicaltrials.gov/large-docs/79/NCT04635579/ICF_002.pdf